CLINICAL TRIAL: NCT01658761
Title: Surgical Outcome of Vitrectomy for Myopic Traction Maculopathy in Highly Myopic Eyes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Principal Investigator, Makoto Inoue, Assosiate professor of Ophthalmology, Kyorin University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KyorinEye008; Myopic maculopathy
Record Dates: First submitted 2012-07-28; First posted 2012-08-07 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Maculopathy; High Myopia; Surgery
Keywords: Myopic traction maculopathy; vitrectomy; internal limiting membrane; Retrospective, case control study
MeSH Terms: conditions — Macular Degeneration | interventions — Vitrectomy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Myopic traction maculopathy (Experimental): The 71 eyes of 64 patients (14 men and 50 women) with myopic traction maculopathy in highly myopic eyes (refractive errors ≤-8.0 diopters and axial length ≥26.0 mm) who underwent vitrectomy were retrospectively reviewed.
  Interventions: Procedure: vitrectomy

INTERVENTIONS:
Procedure: vitrectomy — Surgery
  Other Names: Myopic traction maculopathy in highly myopic eyes

SUMMARY:
Surgical outcome of vitrectomy for myopic traction maculopathy in highly myopic eyes was evaluated in each stage. Efficacy of internal limiting membrane was also evaluated whether it may improve visual outcome.

DETAILED DESCRIPTION:
Surgical outcome of vitrectomy for myopic traction maculopathy in highly myopic eyes was evaluated in each stage of macular retinischisis, foveal detachment, or macular hole. Efficacy of internal limiting membrane was also evaluated whether it may improve visual outcome.

ELIGIBILITY:
Inclusion Criteria:

* Eyes with myopic traction maculopathy in highly myopic eyes with refractive errors ≤ -8.0 diopters and axial length ≥ 26.0 mm who underwent vitrectomy

Exclusion Criteria:

* Eyes with follow-up less than a year

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 1998-09; Primary Completion 2011-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Visual acuity | One year
  Preoperative and postoperative visual acuity

SECONDARY OUTCOMES:
Optical coherence tomography | One year
  Anatomical retinal images by optical cohernce tomography

CONTACTS AND LOCATIONS:
Overall Officials: Makoto Inoue, MD, Principal Investigator — Kyorin Eye Center
Locations (1):
- Kyorin Eye Center, Mitaka, Tokyo, Japan